CLINICAL TRIAL: NCT04916561
Title: Detection of Covid-19 in Tissue Samples of Orthopedic Origin: a Prospective Cohort Study
Brief Title: Detection of Covid-19 in Tissue Samples of Orthopedic Origin
Status: Completed | Type: Observational
Sponsor: Centre de l'arthrose, Paris (Other)
Collaborators: Beaujon Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CovidOS_2020
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: COVID
MeSH Terms: interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: RT-PCR — Detection of Covid-19 in bone, articular fluid and muscle samples using RT-PCR

SUMMARY:
Background The presence of the Covid-19 virus has been detected in tissues of various origins: nasopharyngeal swabs, sputum, bronchoalveolar fluid, blood, stool and anal swabs. However, it does not appear that the virus is excreted in the urine. The REACTing group (Research & Action Emerging Infectious Diseases) has demonstrated the presence of the virus in the conjunctiva and pleural fluid. This detection was made possible by carrying out quantitative, real-time RT-PCR and sequencing of the viral genes, which are currently the benchmark for the diagnosis of COVID-19. However, it is not known at this time whether the Covid-19 virus is present in joint fluid or in bone.

However, some viruses have a particular bone tropism (Parvovirus B19, HHV6); others have joint tropism (parvovirus B19, HBV, HCV, rubella, HIV, HTLV-1). The presence in "orthopedic" tissues of the various coronaviruses (MERS, SARS, etc.) has never been evaluated in the past. However, cases of pulmonary contamination by coronavirus after bone marrow transplantation have been reported in the literature. A potential location at these levels could cause problems of different kinds.

Rationale First, and concretely, a possible direct transmission by these tissues. The current English and Spanish national recommendations in orthopedics show a controversy as to the risk of intraoperative contamination during medical procedures generating aerosols, in particular those involving instruments at high speed (saw blade, reamer, drill). This transmission could also be a problem during bone marrow transplants, from the iliac crests, for example.

Second, but hypothetically, Covid-19 could become quiescent at the level of the myelo-hematopoietic niches and reactivate at a distance, which could then explain the current interrogation on "absence of immunity" and cases of early revival in patients considered cured. This hypothesis is all the more likely since, always by analogy with Parvovirus B19 or HHV6, a recent alert on cases of myocarditis in children has been issued in Parisian pediatric hospitals and that treatment with tocilizumab, which blocks the action Interleukin 6 receptors, and initially used for joint manifestations of rheumatoid arthritis, appear promising.

DETAILED DESCRIPTION:
* Objective: The objective is to determine if Covid-19 is present in bone and joint tissue from operative parts, extracted during routine procedures, in patients diagnosed with Covid + before the procedure.
* Methods: Sample form orthopedics procedure that is usually collected will be analysed for the detection of Covid-19
* Hypothesis: The presence of the virus in the blood suggests a variable amount of presence in the bone tissues, and to a lesser extent articular, of the weakness of their poor vascularity.

Nevertheless, if this is confirmed, understanding of the natural history of the disease would be greatly improved.In the absence of a virus, this would end the controversy about the possibility of contamination by accident from exposure to the block and modify the national recommendations for good orthopedic practices.

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for traumatology or orthopedics procedure.
* > 18 years-old with no upper age limit
* diagnosed Covid+ using RT-PCR during the past one month

Exclusion Criteria:

* Pregnant or lactating women or in age to procreate without contraceptive treatment
* History of mental illness or neurological deficit or adults lacking capacity to consent for themselves
* Prisoners or young offenders
* Persons who might not adequately understand verbal explanations or written information given in French, or who have special communication needs
* Subjects having been or being under an infectious or oncological intercurrent disorder
* Heart failure with risk of exercise angina or comorbidity(ies) significantly affecting patient function
* Any participants who are involved in current research or have recently been involved in any research prior to recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients planned to undergo orthopedic or trauma surgery, and having had a nasopharyngeal sample in their clinical history which was recognized as positive by RT-PCR.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
positive detection rate | immediately after surgery
  rate of patients with possible detection of the virus in an orthopedic sample

SECONDARY OUTCOMES:
viremia | immediately after surgery
  virus detection levels in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Cedric Maillot, MD, Principal Investigator — APHP
Locations (1):
- Université de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will only be done on request and after acceptance of the sponsor's scientific committee if the request is properly justified